CLINICAL TRIAL: NCT01196286
Title: Multifamily Psychoeducation and Cognitive Remediation for Recent-Onset Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Institute for Mental Health Research (Unknown)
Responsible Party: Principal Investigator, Nicholas Breitborde, Assistant Professor, Department of Psychiatry, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-BN-07
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Recent-Onset Psychosis; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder With Psychotic Features; Major Depression With Psychotic Features; Psychotic Disorder Not Otherwise Specified (NOS)
Keywords: First-episode psychosis; cognitive remediation; family psychoeducation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MFG and CR (Experimental): Subjects provided with both multifamily psychoeducation (MFG) and cognitive remediation (CR)
  Interventions: Behavioral: Multifamily Group Psychoeducation (MFG); Behavioral: Cognitive Remediation (CR)
- MFG (Active Comparator): Subjects provided with only multifamily group psychoeducation (MFG)
  Interventions: Behavioral: Multifamily Group Psychoeducation (MFG)

INTERVENTIONS:
Behavioral: Multifamily Group Psychoeducation (MFG) — Participation in multifamily psychoeducation comprised of (i) three individual sessions with family and individual with psychosis, (ii) one psychoeducational workshop, and (iiI) twice monthly multifamily meetings to complete structured problem-solving activity
Behavioral: Cognitive Remediation (CR) — Computer exercises designed to improve cognitive functioning (3hr/wk).
  Arms: MFG and CR

SUMMARY:
The goal of this study is to determine whether pairing multifamily group psychoeducation with cognitive remediation may facilitate improved outcomes among individuals with recent-onset psychosis.

ELIGIBILITY:
Inclusion Criteria (Individual with Recent-Onset Psychosis):

* Diagnosis of a non-substance induced psychotic disorder per DSM-IV-TR criteria determined using the Structured Clinical Interview for the DSM-IV.
* Age between 18-35
* Willing to participate in interventions at University of Arizona Medical Center, South Campus
* Willing to complete research assessments
* Duration of psychotic symptoms of less than 5 years determined using the Symptom Onset in Schizophrenia inventory
* Able to provide informed consent
* Fluent in English
* Must have a family caregiver who is willing to participate in the study
* Willing to allow videotaping of multifamily group therapy sessions.
* No evidence of mental retardation as defined as never having qualified to receive services from the Arizona Department of Economic Security, Division of Developmental Disabilities.

Exclusion Criteria (Individual with Recent-Onset Psychosis):

* Failure to meet inclusion criteria

Inclusion Criteria (Caregiving Relative of Individual with Recent-Onset Psychosis):

* Must be someone that the individual with recent-onset psychosis identifies as providing support and care to the individual with recent-onset psychosis. Does not need to be a biological relative.
* Must spend considerable time with the individual with recent-onset psychosis as defined at 10 hours or more of direct contact per week.
* Willing to participate in participate in family intervention at University of Arizona Medical Center, South Campus for 2 years
* Willing to complete research assessments
* Able to provide informed consent
* Fluent in English
* Willing to allow videotaping of multifamily group sessions.

Exclusion Criteria (Caregiving Relative of Individual with Recent-Onset Psychosis):

* Failure to meet inclusion criteria

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Psychotic Symptoms/Relapse Assessed Once Per Week | 9 months

SECONDARY OUTCOMES:
Depression, Anxiety, Emotional Awareness, Cognitive Functioning, Problem-Solving Ability, Quality of Life, Social Functioning, Service Utilization | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Breitborde, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Background] Breitborde NJ, Woods SW, Srihari VH. Multifamily psychoeducation for first-episode psychosis: a cost-effectiveness analysis. Psychiatr Serv. 2009 Nov;60(11):1477-83. doi: 10.1176/ps.2009.60.11.1477. PMID 19880465
- [Background] Rubinstein E, Breitborde NJ, Jenkins JH. Anthropological intervention early in psychosis. Early Interv Psychiatry. 2010 May;4(2):108-10. doi: 10.1111/j.1751-7893.2010.00175.x. No abstract available. PMID 20536965
- [Background] Breitborde NJ, Srihari VH, Pollard JM, Addington DN, Woods SW. Mediators and moderators in early intervention research. Early Interv Psychiatry. 2010 May;4(2):143-52. doi: 10.1111/j.1751-7893.2010.00177.x. PMID 20536970
- [Derived] Breitborde NJ, Moreno FA, Mai-Dixon N, Peterson R, Durst L, Bernstein B, Byreddy S, McFarlane WR. Multifamily group psychoeducation and cognitive remediation for first-episode psychosis: a randomized controlled trial. BMC Psychiatry. 2011 Jan 12;11:9. doi: 10.1186/1471-244X-11-9. PMID 21226941